CLINICAL TRIAL: NCT05451953
Title: Apneic Oxygenation to Prevent Oxygen Desaturation During Intubation in the NICU
Brief Title: Providing Oxygen During Intubation in the NICU Trial
Acronym: POINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Elizabeth Foglia, Assistant Professor of Pediatrics, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-017190; R21HD103927 (NIH)
Record Dates: First submitted 2022-06-07; First posted 2022-07-11 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Neonatal Respiratory Failure; Tracheal Intubation Morbidity
Keywords: Apneic Oxygenation; Tracheal Intubation; Neonate
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallel group open-label randomized controlled trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apneic Oxygenation (Experimental)
  Interventions: Procedure: Apneic Oxygenation
- Standard of Care (Active Comparator)
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Procedure: Apneic Oxygenation — Nasal cannula at a rate of 6L/min with 100% FiO2 during laryngoscopy and intubation attempt(s)
  Arms: Apneic Oxygenation
Procedure: Standard of Care — No respiratory support during laryngoscopy and intubation attempt(s) (current standard of care)
  Arms: Standard of Care

SUMMARY:
Tracheal intubation in the NICU is frequently complicated by severe oxygen desaturation. Apneic oxygenation, a method of applying free flowing oxygen via nasal cannula to apneic patients undergoing intubation, prevents or delays oxygen desaturation during intubation in adults and older children. We propose to enroll patients at two sites (Hospital of the University of Pennsylvania and Children's Hospital of Philadelphia) in a randomized trial in infants undergoing intubation in the NICU to determine if apneic oxygenation, compared with no respiratory support or oxygen during laryngoscopy and intubation attempts (standard care), reduces the magnitude of oxygen desaturation during tracheal intubation encounters.

ELIGIBILITY:
Inclusion Criteria:

1. Infants ≥28 weeks corrected gestational age
2. Undergoing intubation in the NICU
3. Pre-medication (including paralytic) administered

Exclusion Criteria:

1. Critical Airway or Airway Anomaly
2. Unstable hemodynamics (i.e. active resuscitation)
3. Unable to achieve SpO2 ≥90% prior to intubation attempt
4. Intubation performed by Non-NICU provider (i.e. anesthesiology or ENT)
5. Unrepaired congenital diagrammatic hernia
6. Tracheal esophageal fistula within 2 weeks of repair
7. Tracheostomy
8. Previous enrollment in the trial
9. Nasal intubation
10. COVID person under investigation (PUI) or COVID positive
11. Cyanotic heart disease
12. Receiving Extracorporeal Membrane Oxygenation support
13. Conjoined twins

Ages: 0 Days to 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary Clinical Outcome: Change in Oxygen Saturation (SpO2) | During intubation procedure
  Difference between highest SpO2 immediately prior to first intubation attempt and lowest SpO2 during the intubation encounter.

SECONDARY OUTCOMES:
Secondary Clinical Outcome: Severe oxygen desaturation | During intubation procedure
  ≥20% decline in SpO2
Secondary Clinical Outcome: SpO2<80% | During intubation procedure
  SpO2<80% at any point
Secondary Clinical Outcome: Time to SpO2 <80% | During intubation procedure
  Time to SpO2 <80% from facemask removal
Secondary Clinical Outcome: intubation success | During intubation procedure
  First intubation attempt success
Secondary Clinical Outcome: Number of intubation attempts | During intubation procedure
  Total number of intubation attempts
Secondary Clinical Outcome: Duration of intubation attempts | During intubation procedure
  Duration of each intubation attempt
Secondary Clinical Outcome: Change in pulse rate | During intubation procedure
  Difference between highest and lowest pulse rate
Secondary Clinical Outcome: pH | Three hours after intubation
  First blood gas pH
Secondary Clinical Outcome: pCO2 | Three hours after intubation
  First blood gas pCO2
Secondary Clinical Outcome: PaO2 | Three hours after intubation
  First blood gas PaO2 (for infants with indwelling arterial lines)
Feasibility Outcome: AO fidelity | During the intubation procedure
  Proportion subjects allocated to AO successfully provided the AO intervention
Feasibility Outcome: Protocol deviations | During intubation procedure
  Number of protocol deviations and violations
Feasibility Outcome: Screening | Through study completion, an average of 18 months.
  Proportion of intubated infants successfully screened in advance
Feasibility Outcome: Recruitment | Through study completion, an average of 18 months.
  Rates of informed consent
Feasibility Outcome: Randomization | Through study completion, an average of 18 months.
  Proportion of consented infants who were randomized

OTHER OUTCOMES:
Safety Outcome: Cardiopulmonary resuscitation | During or within 1 hour of procedure
  Chest compressions with or without epinephrine
Safety Outcome: Air Leaks | Within 24 hours of procedure
  New pneumothorax
Safety Outcome: Nasal Trauma | Within 24 hours of procedure
  New nasal trauma
Safety Outcome: adverse Tracheal Intubation Adverse Events | During Intubation Procedure
  Tracheal Intubation Adverse Events, per NEAR4NEOS definitions
Safety Outcome: Duration of time with 100% SpO2 | During Intubation Procedure
  Duration of time with SpO2=100%

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Foglia, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will make data available after study completion and in accordance with NIH policies. Our data will only be provided to those investigators who agree to adhere to a signed research data use agreement. The execution of the agreement will require approval by the institution's IRB or demonstration of IRB exemption per institutional policy. The data and the associated documentation will be available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and does not identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, ICF
Time Frame: After study completion.
Access Criteria: Data use agreement in place prior to data sharing.

REFERENCES:
- [Background] Di Fiore JM, Poets CF, Gauda E, Martin RJ, MacFarlane P. Cardiorespiratory events in preterm infants: interventions and consequences. J Perinatol. 2016 Apr;36(4):251-8. doi: 10.1038/jp.2015.165. Epub 2015 Nov 19. PMID 26583943
- [Background] Drianovski P. [The problem of radiation resistance in birds]. Vet Med Nauki. 1974;11(4):91-7. No abstract available. Bulgarian. PMID 4428609
- [Background] Whalley ET, Wahl M, Sampaio CA. Angiotensin-converting enzyme, bradykinin, angiotensin, and cerebral vessel reactivity. Hypertension. 1983 Nov-Dec;5(6 Pt 3):V34-7. doi: 10.1161/01.hyp.5.6_pt_3.v34. PMID 6317557
- [Background] Poets CF, Roberts RS, Schmidt B, Whyte RK, Asztalos EV, Bader D, Bairam A, Moddemann D, Peliowski A, Rabi Y, Solimano A, Nelson H; Canadian Oxygen Trial Investigators. Association Between Intermittent Hypoxemia or Bradycardia and Late Death or Disability in Extremely Preterm Infants. JAMA. 2015 Aug 11;314(6):595-603. doi: 10.1001/jama.2015.8841. PMID 26262797
- [Background] Kumar P, Denson SE, Mancuso TJ; Committee on Fetus and Newborn, Section on Anesthesiology and Pain Medicine. Premedication for nonemergency endotracheal intubation in the neonate. Pediatrics. 2010 Mar;125(3):608-15. doi: 10.1542/peds.2009-2863. Epub 2010 Feb 22. PMID 20176672
- [Background] Grude O, Solli HJ, Andersen C, Oveland NP. Effect of nasal or nasopharyngeal apneic oxygenation on desaturation during induction of anesthesia and endotracheal intubation in the operating room: A narrative review of randomized controlled trials. J Clin Anesth. 2018 Dec;51:1-7. doi: 10.1016/j.jclinane.2018.07.002. Epub 2018 Jul 18. PMID 30029021
- [Background] Steiner JW, Sessler DI, Makarova N, Mascha EJ, Olomu PN, Zhong JW, Setiawan CT, Handy AE, Kravitz BN, Szmuk P. Use of deep laryngeal oxygen insufflation during laryngoscopy in children: a randomized clinical trial. Br J Anaesth. 2016 Sep;117(3):350-7. doi: 10.1093/bja/aew186. Epub 2016 Jul 27. PMID 27466252
- [Background] Windpassinger M, Plattner O, Gemeiner J, Roder G, Baumann A, Zimmerman NM, Sessler DI. Pharyngeal Oxygen Insufflation During AirTraq Laryngoscopy Slows Arterial Desaturation in Infants and Small Children. Anesth Analg. 2016 Apr;122(4):1153-7. doi: 10.1213/ANE.0000000000001189. PMID 26991620
- [Background] Humphreys S, Lee-Archer P, Reyne G, Long D, Williams T, Schibler A. Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) in children: a randomized controlled trial. Br J Anaesth. 2017 Feb;118(2):232-238. doi: 10.1093/bja/aew401. PMID 28100527
- [Background] Napolitano N, Laverriere EK, Craig N, Snyder M, Thompson A, Davis D, Nett S, Branca A, Harwayne-Gidansky I, Sanders R Jr, Shults J, Nadkarni V, Nishisaki A; National Emergency Airway Registry for Children (NEAR4KIDS) and Pediatric Acute Lung Injury and Sepsis Investigators (PALISI). Apneic Oxygenation As a Quality Improvement Intervention in an Academic PICU. Pediatr Crit Care Med. 2019 Dec;20(12):e531-e537. doi: 10.1097/PCC.0000000000002123. PMID 31568243
- [Background] Long E, Cincotta DR, Grindlay J, Sabato S, Fauteux-Lamarre E, Beckerman D, Carroll T, Quinn N. A quality improvement initiative to increase the safety of pediatric emergency airway management. Paediatr Anaesth. 2017 Dec;27(12):1271-1277. doi: 10.1111/pan.13275. Epub 2017 Oct 24. PMID 29063722
- [Background] Vukovic AA, Hanson HR, Murphy SL, Mercurio D, Sheedy CA, Arnold DH. Apneic oxygenation reduces hypoxemia during endotracheal intubation in the pediatric emergency department. Am J Emerg Med. 2019 Jan;37(1):27-32. doi: 10.1016/j.ajem.2018.04.039. Epub 2018 Apr 18. PMID 29699900
- [Background] Nishisaki A, Turner DA, Brown CA 3rd, Walls RM, Nadkarni VM; National Emergency Airway Registry for Children (NEAR4KIDS); Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. A National Emergency Airway Registry for children: landscape of tracheal intubation in 15 PICUs. Crit Care Med. 2013 Mar;41(3):874-85. doi: 10.1097/CCM.0b013e3182746736. PMID 23328260
- [Background] Li S, Hsieh TC, Rehder KJ, Nett S, Kamat P, Napolitano N, Turner DA, Adu-Darko M, Jarvis JD, Krawiec C, Derbyshire AT, Meyer K, Giuliano JS Jr, Tala J, Tarquinio K, Ruppe MD, Sanders RC Jr, Pinto M, Howell JD, Parker MM, Nuthall G, Shepherd M, Emeriaud G, Nagai Y, Saito O, Lee JH, Simon DW, Orioles A, Walson K, Vanderford P, Shenoi A, Lee A, Bird GL, Miksa M, Graciano AL, Bain J, Skippen PW, Polikoff LA, Nadkarni V, Nishisaki A; for National Emergency Airway Registry for Children (NEAR4KIDS) and Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Frequency of Desaturation and Association With Hemodynamic Adverse Events During Tracheal Intubations in PICUs. Pediatr Crit Care Med. 2018 Jan;19(1):e41-e50. doi: 10.1097/PCC.0000000000001384. PMID 29210925
- [Background] Brown CA 3rd, Bair AE, Pallin DJ, Walls RM; NEAR III Investigators. Techniques, success, and adverse events of emergency department adult intubations. Ann Emerg Med. 2015 Apr;65(4):363-370.e1. doi: 10.1016/j.annemergmed.2014.10.036. Epub 2014 Dec 20. PMID 25533140
- [Background] Neumann RP, von Ungern-Sternberg BS. The neonatal lung--physiology and ventilation. Paediatr Anaesth. 2014 Jan;24(1):10-21. doi: 10.1111/pan.12280. Epub 2013 Oct 24. PMID 24152199
- [Background] Patel R, Lenczyk M, Hannallah RS, McGill WA. Age and the onset of desaturation in apnoeic children. Can J Anaesth. 1994 Sep;41(9):771-4. doi: 10.1007/BF03011582. PMID 7954992
- [Background] Haubner LY, Barry JS, Johnston LC, Soghier L, Tatum PM, Kessler D, Downes K, Auerbach M. Neonatal intubation performance: room for improvement in tertiary neonatal intensive care units. Resuscitation. 2013 Oct;84(10):1359-64. doi: 10.1016/j.resuscitation.2013.03.014. Epub 2013 Apr 3. PMID 23562374
- [Background] Durrmeyer X, Breinig S, Claris O, Tourneux P, Alexandre C, Saliba E, Beuchee A, Jung C, Levy C, Marchand-Martin L, Marcoux MO, Dechartres A, Danan C; PRETTINEO Research Group. Effect of Atropine With Propofol vs Atropine With Atracurium and Sufentanil on Oxygen Desaturation in Neonates Requiring Nonemergency Intubation: A Randomized Clinical Trial. JAMA. 2018 May 1;319(17):1790-1801. doi: 10.1001/jama.2018.3708. PMID 29715354
- [Background] Roberts KD, Leone TA, Edwards WH, Rich WD, Finer NN. Premedication for nonemergent neonatal intubations: a randomized, controlled trial comparing atropine and fentanyl to atropine, fentanyl, and mivacurium. Pediatrics. 2006 Oct;118(4):1583-91. doi: 10.1542/peds.2006-0590. PMID 17015550
- [Background] O'Shea JE, Thio M, Kamlin CO, McGrory L, Wong C, John J, Roberts C, Kuschel C, Davis PG. Videolaryngoscopy to Teach Neonatal Intubation: A Randomized Trial. Pediatrics. 2015 Nov;136(5):912-9. doi: 10.1542/peds.2015-1028. Epub 2015 Oct 19. PMID 26482669
- [Background] Moussa A, Luangxay Y, Tremblay S, Lavoie J, Aube G, Savoie E, Lachance C. Videolaryngoscope for Teaching Neonatal Endotracheal Intubation: A Randomized Controlled Trial. Pediatrics. 2016 Mar;137(3):e20152156. doi: 10.1542/peds.2015-2156. Epub 2016 Feb 12. PMID 26908701
- [Background] Oliveira J E Silva L, Cabrera D, Barrionuevo P, Johnson RL, Erwin PJ, Murad MH, Bellolio MF. Effectiveness of Apneic Oxygenation During Intubation: A Systematic Review and Meta-Analysis. Ann Emerg Med. 2017 Oct;70(4):483-494.e11. doi: 10.1016/j.annemergmed.2017.05.001. Epub 2017 Jul 14. PMID 28712606
- [Background] Cummings JJ, Polin RA, COMMITTEE ON FETUS AND NEWBORN. Oxygen Targeting in Extremely Low Birth Weight Infants. Pediatrics. 2016;138(2):e20161576. Pediatrics. 2016 Dec;138(6):e20162904. doi: 10.1542/peds.2016-2904. No abstract available. PMID 27940728
- [Background] Dempsey EM, Al Hazzani F, Faucher D, Barrington KJ. Facilitation of neonatal endotracheal intubation with mivacurium and fentanyl in the neonatal intensive care unit. Arch Dis Child Fetal Neonatal Ed. 2006 Jul;91(4):F279-82. doi: 10.1136/adc.2005.087213. Epub 2006 Feb 7. PMID 16464937
- [Background] Johnston L, Sawyer T, Nishisaki A, Whitfill T, Ades A, French H, Glass K, Dadiz R, Bruno C, Levit O, Gangadharan S, Scherzer D, Moussa A, Auerbach M; INSPIRE Research Network. Neonatal Intubation Competency Assessment Tool: Development and Validation. Acad Pediatr. 2019 Mar;19(2):157-164. doi: 10.1016/j.acap.2018.07.008. Epub 2018 Aug 11. PMID 30103050
- [Background] Venkatesh V, Ponnusamy V, Anandaraj J, Chaudhary R, Malviya M, Clarke P, Arasu A, Curley A. Endotracheal intubation in a neonatal population remains associated with a high risk of adverse events. Eur J Pediatr. 2011 Feb;170(2):223-7. doi: 10.1007/s00431-010-1290-8. Epub 2010 Sep 15. PMID 20842378
- [Background] Gupta S, Donn SM. Continuous positive airway pressure: Physiology and comparison of devices. Semin Fetal Neonatal Med. 2016 Jun;21(3):204-11. doi: 10.1016/j.siny.2016.02.009. Epub 2016 Mar 3. PMID 26948884
- [Background] Roberts CT, Owen LS, Manley BJ, Davis PG; Australian & New Zealand Neonatal Network (ANZNN). High-flow support in very preterm infants in Australia and New Zealand. Arch Dis Child Fetal Neonatal Ed. 2016 Sep;101(5):F401-3. doi: 10.1136/archdischild-2015-309328. Epub 2015 Dec 17. PMID 26678879
- [Background] Roberts CT, Owen LS, Manley BJ, Froisland DH, Donath SM, Dalziel KM, Pritchard MA, Cartwright DW, Collins CL, Malhotra A, Davis PG; HIPSTER Trial Investigators. Nasal High-Flow Therapy for Primary Respiratory Support in Preterm Infants. N Engl J Med. 2016 Sep 22;375(12):1142-51. doi: 10.1056/NEJMoa1603694. PMID 27653564
- [Background] Yoder BA, Stoddard RA, Li M, King J, Dirnberger DR, Abbasi S. Heated, humidified high-flow nasal cannula versus nasal CPAP for respiratory support in neonates. Pediatrics. 2013 May;131(5):e1482-90. doi: 10.1542/peds.2012-2742. Epub 2013 Apr 22. PMID 23610207
- [Background] Bresesti I, Zivanovic S, Ives KN, Lista G, Roehr CC. National surveys of UK and Italian neonatal units highlighted significant differences in the use of non-invasive respiratory support. Acta Paediatr. 2019 May;108(5):865-869. doi: 10.1111/apa.14611. Epub 2018 Nov 13. PMID 30307647
- [Background] Wilkinson DJ, Andersen CC, Smith K, Holberton J. Pharyngeal pressure with high-flow nasal cannulae in premature infants. J Perinatol. 2008 Jan;28(1):42-7. doi: 10.1038/sj.jp.7211879. Epub 2007 Nov 8. PMID 17989697
- [Background] Nielsen KR, Ellington LE, Gray AJ, Stanberry LI, Smith LS, DiBlasi RM. Effect of High-Flow Nasal Cannula on Expiratory Pressure and Ventilation in Infant, Pediatric, and Adult Models. Respir Care. 2018 Feb;63(2):147-157. doi: 10.4187/respcare.05728. Epub 2017 Oct 24. PMID 29066588
- [Background] Lee JH, Turner DA, Kamat P, Nett S, Shults J, Nadkarni VM, Nishisaki A; Pediatric Acute Lung Injury and Sepsis Investigators (PALISI); National Emergency Airway Registry for Children (NEAR4KIDS). The number of tracheal intubation attempts matters! A prospective multi-institutional pediatric observational study. BMC Pediatr. 2016 Apr 29;16:58. doi: 10.1186/s12887-016-0593-y. PMID 27130327
- [Derived] Herrick HM, O'Reilly M, Lee S, Wildenhain P, Napolitano N, Shults J, Nishisaki A, Foglia EE. Providing Oxygen during Intubation in the NICU Trial (POINT): study protocol for a randomised controlled trial in the neonatal intensive care unit in the USA. BMJ Open. 2023 Apr 13;13(4):e073400. doi: 10.1136/bmjopen-2023-073400. PMID 37055198